CLINICAL TRIAL: NCT04112173
Title: Fall-recovery Training for Those With Chronic Stroke and Low Falls Self-efficacy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study activity has initially suspended due to COVID-19 restrictions, but it will not resume due to the confounding influence of the pandemic on the study outcomes. The feasibility of the study protocol is limited with restrictions from the pandemic.
Sponsor: University of Delaware (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Jeremy Crenshaw, Principal Investigator, University of Delaware
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1490979-1; U54GM104941 (NIH)
Record Dates: First submitted 2019-09-16; First posted 2019-10-02 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: balance; self-efficacy; exercise; postural control
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: single-group, observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perturbation-Based Balance Training (Experimental): perturbation-based balance training
  Interventions: Behavioral: perturbation-based fall-recovery training

INTERVENTIONS:
Behavioral: perturbation-based fall-recovery training — Participants will attempt to recover from treadmill-induced balance perturbations as they walk or stand. The size of the perturbations is progressively challenging and dependent upon participant performance.
  Other Names: balance training

SUMMARY:
Chronic stroke is the leading cause of long-term disability in the United States. Post-stroke health is negatively impacted by two interrelated factors-a substantial risk of falls and limited walking activity. The risk of falling is a barrier to walking activity, with falls self-efficacy mediating the relationship between impaired physical capacity and limited activity. The ability to recover from a fall (i.e. arrest a fall before impact) is a logical, yet untested rehabilitation target to enable walking activity through sustained benefits to falls self-efficacy. Our aim is to demonstrate that fall-recovery training is feasible in stroke survivors with low falls self-efficacy. Five participants will undergo an adapted version of fall-recovery training. We will gather evidence of the implementation, adaptation, and limited efficacy of this intervention in affecting falls self-efficacy and walking activity.

DETAILED DESCRIPTION:
The study aim is to demonstrate that fall-recovery training is feasible in stroke survivors with low falls self-efficacy. We will gather evidence of the adaptation, implementation, and limited efficacy of our intervention. This aim will be addressed with a single-group, interventional study. At baseline, fall-recovery ability will be determined from stepping thresholds in response to treadmill-delivered perturbations. Falls self-efficacy will be determined from questionnaires. Walking activity will be recorded using step counters (StepWatchTM). After three weeks of a non-active control period, we will repeat assessments. Then, participants will attend six training sessions consisting of anterior, posterior, and lateral perturbations. After training, we will repeat all assessments of balance, self-efficacy, and walking activity. We will recruit five participants with chronic stroke (i.e. >6 months after stroke). Falls self-efficacy is recorded upon registry enrollment, allowing us to recruit to our study needs. All participants must have an Activities-Specific Balance Confidence (ABC) score less than 68. Upon enrollment, the Fugl-Meyer Lower Extremity assessment and Stroke Impact Scale will be administered. Fall-recovery ability will be quantified from anterior, posterior, and lateral single-stepping thresholds. Participants will be outfitted with a harness attached to an overhead rail. As they stand on a computer-controlled treadmill (ActiveStep®, Simbex), participants will be instructed to not step in response to rapid belt translations. For each opposing pair of thresholds, a progressively challenging series of perturbations will be delivered. Thresholds are defined as the perturbation magnitudes that consistently elicit one step. Falls self-efficacy will be quantified from the ABC scale and the Falls Efficacy Scale (FES). Walking activity will be quantified as average daily steps, recorded in five-second intervals for one week by a StepWatchTM monitor on the non-paretic ankle.

Our fall-recovery training consists of 6 sessions over 3-4 weeks, each consisting of the following 5-minute series:

* Standing perturbations that induce a forward fall, necessitating multiple steps to regain stability. Separate series will focus on paretic and non-paretic steps. Participants will be instructed to "try not to fall".
* Standing perturbations that induce a backwards fall. Instructions will be to recover in a single step. This constraint is added because, unlike the multiple-step response of trip recoveries, slip recovery is dictated by first-step features. Separate series will focus on initial steps with the paretic or non-paretic limb.
* Standing perturbations that induce a lateral fall, delivered as participants stand facing the side of the treadmill. Participants will be instructed to "try not to fall". We will apply left and right perturbations large enough to elicit a step.
* Also, we will apply anterior and posterior perturbations as the participants walk. Our treadmill is equipped to deliver perturbations timed relative to foot strikes during gait.

The training intensity, as determined by the perturbation size and, if applicable, gait speed, will be small at first, progressing to more challenging levels dependent upon participant performance, safety, and comfort.

As per feasibility-study guidelines, we will gather evidence of adaptation, implementation, and limited efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older
* Participants must have had a single stroke of non-cerebellar origin, occurring six or more months prior to study enrollment.
* An Activities-Specific Balance Confidence (ABC) score less than 68.

Exclusion Criteria:

* More than one stroke
* Acute illness at the time of functional assessment or training
* Body mass greater than 136 kg (300 lbs) to ensure that the treadmill accelerates accurately
* Lower extremity joint replacement or shoulder joint replacement within a year prior to participation
* Dementia
* Parkinson's disease
* A history of back surgery
* A history of neck surgery
* More than one occurrence of back or neck pain in the month prior to participation
* Current back or neck pain at the time of participant enrollment
* Bulging vertebral discs
* Spine, hip, or lower extremity fracture within a year prior to participation
* Open lesions on the lower extremity
* Insulin-dependent diabetes
* Use of a pacemaker
* Use of an ostomy pouch
* Pregnancy
* Osteoporosis
* Doctor recommendation to avoid moderate physical activity or exercise
* Any neural, muscular, or skeletal condition or injury that precludes safe participation in the training or introduces a confounding factor on the study, at the discretion of the clinician or study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant recruited on 2/21/2020 at University of Delaware campus.
Period: Overall Study
Arm/Group | Perturbation-based Balance Training
Started | 1
Completed | 0 (Study halted on 3/13/2020 due to COVID-19 pandemic. Study was terminated without resuming.)
Not Completed | 1
Not completed — Study terminated due to COVID-19 pandemic | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention: perturbation-based balance training
  perturbation-based fall-recovery training: Participants will attempt to recover from treadmill-induced balance perturbations as they walk or stand. The size of the perturbations is progressively challenging and dependent upon participant performance.
Arm/Group | Intervention
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 56 [56 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Balance Confidence [Number; unit: units on a scale] — The Activities- Specific Balance Confidence (ABC) Scale is a self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness.
  Range 0-100 Higher values represent a better outcome.
  units on a scale | 52
Lower Extremity Fugl-Meyer [Number; unit: units on a scale] — The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia
  Scores range from 0-34 Higher values represent a better outcome.
  units on a scale | 20
Stroke Impact Scale [Number; unit: units on a scale] — The stroke impact scale is a self-report questionnaire that evaluates disability and health-related quality of life after stroke.
  Range for each domain (0-100)
  Domain scores are averaged for total score.
  Higher values represent a better outcome.
  units on a scale
    Strength | 12.5
    Memory and Thinking | 83.3
    Emotions | 83.3
    Communication | 64.3
    ADL/IADL | 70
    Mobility | 66.7
    Hand Function | 0
    Participation/Role | 68.8
Anteroposterior stepping thresholds [Number; unit: m/s^2] — As participants stand on a computer-controlled treadmill, sudden belt accelerations perturb balance. Perturbations are delivered in forward and backward directions, and participants are instructed to not step. The size of the perturbations is increased until the participant steps in response to the movement. Thresholds are defined as the acceleration of the treadmill belt (in units of m/s^2) that consistently elicited an anterior or posterior step.
  m/s^2
    Anterior | 1
    Posterior | 2.5
Falls Efficacy Scale [Number; unit: units on a scale] — A 16-item self-administered questionnaire designed to assess fear of falling
  Range: 16-64
  Lower values represent a better outcome.
  units on a scale | 38

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Ending Participation
Description: The number of participants who end participation due to adverse events
Time Frame: 6 months
Population: The study was terminated prior to reaching the pre-specified time frame for recording this data. This outcome measure was not recorded.
Arm/Group | Intervention
Number analyzed (Participants) | 0

2. Primary Outcome: Activities Specific Balance Confidence Questionnaire Score.
Description: Balance confidence, as measured by the Activities Specific Balance Confidence questionnaire. Scores range from 0 to 100, and represent the average rating of each question. Higher scores indicate more confidence.
  Range 0-100
  Higher values represent a better outcome.
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Intervention
Number analyzed (Participants) | 0

3. Primary Outcome: Falls Self-Efficacy Scale Score
Description: Falls Self-Efficacy, as measured by the Falls Self-Efficacy Scale. Scores are totaled, ranging from 16-64, with higher scores representing worse self-efficacy.
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Intervention
Number analyzed (Participants) | 0

4. Primary Outcome: Walking Activity
Description: Average steps/day, as measured by a step monitor
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Intervention
Number analyzed (Participants) | 0

5. Secondary Outcome: Stepping Threshold Assessment of Reactive Balance
Description: Stepping thresholds are the treadmill-induced, standing perturbation magnitudes that elicit anterior, posterior, or lateral steps. These thresholds are determined from a series of progressively challenging perturbations, delivered as participants stand on a computer-controlled treadmill. The thresholds are the size of the perturbation (measured as acceleration) that results in a step for four trial. Participants are instructed to try not to step. One progression consists of forward and backward perturbations to determine anterior and posterior thresholds. A second progression is done with participants facing the side of the treadmill, with the progression identifying left and right stepping thresholds. Anterior, posterior, left, and right thresholds are considered independently (i.e. not averaged or summed).
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Intervention
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 month (from study start date: February 21, 2020 to the day the study was halted: March 13, 2020).
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was halted due to the COVID-10 pandemic after one participant was enrolled and completed baseline assessments. The study did not resume and participation was terminated by the investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT04112173/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT04112173/ICF_001.pdf